CLINICAL TRIAL: NCT07061912
Title: A Study to Evaluate the Performance of INSTI® HIV Self Test When Performed by Unobserved Intended Users in the US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CLS-003A
Record Dates: First submitted 2025-07-08; First posted 2025-07-14 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Human Immunodeficiency Virus I Infection; Human Immunodeficiency Virus II Infection
Keywords: HIV Self Test; INSTI HIV Self Test; At-Home HIV Test

STUDY DESIGN:
Masking Description: As there is a potential for recruiting known HIV subjects, the care providers will be blinded to the subject's status during testing procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Performance (Experimental): INSTI® HIV ST devices are provided to the enrolled participants to conduct the self test using the provided instruction for use, unobserved. The participant records the INSTI® HIV ST results. The operator then enters the room and also interprets the participants self-test, the operator then performs the comparator test to compare the results with the INSTI® HIV ST.
  Interventions: Device: NSTI® HIV Self-Test

INTERVENTIONS:
Device: NSTI® HIV Self-Test — Each participant will be provided with the INSTI® HIV Self-Test(s) and asked to conduct self testing, unobserved. The participant will record their interpretation of the results. Subjects will perform the test without intervention or observation from the operator. The operator will then enter the room and also interpret the subject's self-test results then perform the comparator test. In the event of a discrepant result between the INSTI® HIV ST and comparator test, an additional venous blood sample will be collected from the subject and sent for discrepancy testing

SUMMARY:
The objective of this study is to evaluate the performance of INSTI® HIV Self Test with unobserved intended user population. The purpose of this study is to document if a lay person, unassisted by a healthcare worker, is able to perform the INSTI® HIV Self Test correctly and without significant risk of incorrect results. The study aims to evaluate the clinical performance (i.e., diagnostic sensitivity and specificity) of the INSTI® HIV Self-Test in a lay user population.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the performance of INSTI® HIV Self Test with unobserved intended user population. The purpose of this study is to document if a lay person, unassisted by a healthcare worker, is able to perform the INSTI® HIV Self Test correctly and without significant risk of incorrect results. The study aims to evaluate the clinical performance (i.e., diagnostic sensitivity and specificity) of the INSTI® HIV Self-Test in a lay user population.

The study population will be based on a general all-comers group of subjects. This includes both unknown HIV status and potentially known HIV positive status subjects.

The number of valid positives from the comparator test will be monitored during the course of the study. When the comparator test reaches 10 valid positive results, the INSTI® HIV ST results for the same 10 subjects will be checked to see if they are also valid. If not, additional subjects will be recruited until there are at least 10 valid INSTI® HIV ST results within the comparator valid positive test results. Once the threshold has been reached recruiting will end. For known HIV positive subjects, site(s) will be requested to provide HIV-1/2 viral load and/or CD4 count laboratory results if available. Additionally, known HIV positive subjects on Anti-Retroviral Treatment (ART) should be on medication for less than 12 months.

The study will initially recruit HIV unknown status subjects, at 50% of total enrollment (i.e., 50 out of 100 subjects) if the 10 HIV positives is deemed unattainable then HIV known subjects may be recruited to make up the 10 total HIV positives.

The study is designed to evaluate INSTI® HIV ST performance when used unobserved by non-professional, untrained intended users that are inexperienced in self-testing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Operator/study staff must complete the subject's Enrolment Questionnaire
* Subject to sign and date the Informed Consent Form
* Able to complete the required testing on the allocated testing day(s)
* Able to speak/ read/write English or Spanish
* Willingness to provide the fingerstick blood sample and if necessary, the volume of whole blood collected through venous blood draw (approximately 7 ml)
* Willingness to participate in the study site's standard of care HIV counselling and testing program and receive the study site's standard of care test results
* Unknown HIV Status or known HIV positive status with less than 12 months of ART
* For known HIV positive status subjects, willingness to share ART start date

Exclusion Criteria:

* Has participated in any prior, or concurrent trial of HIV self-tests
* Is a practicing medical healthcare professional (doctor, nurse or HIV Counsellor that performs HIV testing with Rapid Tests)
* Has used a Rapid Diagnostic Test for HIV blood-based self-testing previously
* Has received any experimental HIV vaccine
* Has a bleeding disorder
* Known HIV positive subjects and currently on an Anti-Retroviral Treatment (ART) for 12 months or longer and/or not willing to share ART start date
* Any condition which, in the opinion of the Operator, would make the participant unsuitable or unsafe for enrolment or could interfere with the completion of the assessment, consent form and questionnaire etc. or bias the outcome, i.e., being unable to see / read by forgetting to bring reading glasses, being intoxicated or acute sickness, or visibly distressed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Clinical sensitivity and specificity of the INSTI® HIV Self-Test | 1 month
  * Percent agreement for fingerstick blood between INSTI® HIV ST results obtained and interpreted by the subject and Comparator Test result obtained by the operator. Percent agreement will be calculated for all sites combined.
  * Point estimate for positive percent agreement will be calculated for all subjects.
  * Negative percent agreement values and 95% CIs will be calculated for all subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- bioLytical Laboratories Inc., Richmond, British Columbia, Canada